CLINICAL TRIAL: NCT04087746
Title: Comparison of Aflibercept Versus Ranibizumab in Management of Diabetic Macular Edema
Brief Title: Comparison of Aflibercept Versus Ranibizumab in Management of Diabetic Macular Edema (DME)
Acronym: DME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minia University & SFH
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- AFLIBERCEPT (Active Comparator): Intra-vitreal injection of AFLIBERCEPT
  Interventions: Drug: Aflibercept
- RANIBIZUMAB (Active Comparator): Intra-vitreal injection of RANIBIZUMAB
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Aflibercept — Intra-vitreal injection of AVEGF AFLIBERCEPT in group I
  Other Names: Group1
  Arms: AFLIBERCEPT
Drug: Ranibizumab — Intra-vitreal injection of AVEGF Ranibizumab in group 2
  Other Names: Group 2
  Arms: RANIBIZUMAB

SUMMARY:
Diabetic macular edema (DME) is a sign of diabetic retinopathy that affects central vision. It is also a leading cause of visual decline in younger patients, especially in developing countries like our Arab community. Intra-vitrreal injection of anti-vascular endothelial growth factor (AVEGF) in management of DME had significant improvement in the final logMAR Un-corrected Distant Visual Acuity ( UCDVA) and logMAR Best Corrected Distant Visual Acuity (BCDVA), as well as reduction in the central retinal thickness from baseline measurement.

DETAILED DESCRIPTION:
The investigators randomly assigned four hundreds eyes of diabetic patients with central diabetic macular edema for intra-vitreal injection of AVEGF group I (200 patients eyes) received aflibercept 2.0 mg and group II (200 patients eyes) received ranibizumab 0.3 mg. Injection was at 4 weeks interval according to the used protocol. The primary outcome was measuring the mean change in visual acuity as functional outcome and the secondary outcomes were the mean change in central macular thickness, as anatomical outcome rather than safety and efficacy of those two anti-VEGF drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or 2 diabetes mellitus with central DME clinically as well as documented by optical coherence tomography (OCT) imaging
* The age of the patients at least 20 years old
* Patients not receiving AVEGF injection, at least for one year
* The BCDVA letter score of at least one eye (range, 0 to 115, with higher scores indicating better visual acuity of 90 (Snellen = 20/32) to 40 (Snellen = 20/320) and central DME .

Exclusion Criteria:

* Patients with cataract
* Glaucoma patient
* Previous AVEGF injection in less than one year
* Patients not attending all of the scheduled follow up visits

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
measuring the main change in visual acuity | 2 years
  measuring the main change in visual acuity in logarithm of the minimum angle of resolution (log MAR) using projector chart as functional outcome

SECONDARY OUTCOMES:
the main change in central macular thickness | 2 years
  the main change in central macular thickness in micrometer by using optical coherence tomography (OCT) as anatomical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban AM Elwan, MD, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patients provided informed written consent for their medical information to be included in analysis and for publication.
Supporting Information: ICF
Time Frame: 2 year
Access Criteria: Full PDF